CLINICAL TRIAL: NCT01350167
Title: Screening for Hepatocellular Carcinoma With Triphasic Helical CT vs. US With Alpha-fetoprotein in Patients With Advanced Liver Disease
Brief Title: Screening for Liver Cancer With CT vs. Ultrasound in Patients With Advanced Liver Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Christine Pocha/Staff Physician, Minneapolis VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 3034-A
Record Dates: First submitted 2011-05-03; First posted 2011-05-09 (Estimated); Last update posted 2011-05-24 (Estimated); Status verified 2010-12

CONDITIONS: Cirrhosis; End Stage Liver Disease; Hepatitis C
Keywords: Hepatocellular Carcinoma; Liver Cancer; Ultrasound; Computed Tomography; Alpha fetoprotein; Cirrhosis; Screening; Advanced Liver Disease
MeSH Terms: conditions — Fibrosis; End Stage Liver Disease; Hepatitis C; Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Triphasic CT (Active Comparator): Triphasic CT of the abdomen with and without contrast every 12 months with alpha-fetoprotein every 6 months.
  Interventions: Procedure: Screening
- Ultrasound (Active Comparator): Ultrasound of the upper left quadrant with alpha-fetoprotein testing every 6 months.
  Interventions: Procedure: Screening

INTERVENTIONS:
Procedure: Screening — Triphasic CT of the abdomen with and without contrast every 12 months and alpha-fetoprotein testing every 6 months. Repeated until HCC diagnosed for up to 10 years.
  Ultrasound of the upper left quadrant every 6 months with alpha-fetoprotein testing every 6 months. Repeated until HCC diagnosed for up to 10 years.

SUMMARY:
The purpose of this study is to determine whether ultrasound or CT scanning is more effective at detecting early liver cancer in patients with advanced liver disease.

DETAILED DESCRIPTION:
Most cases of hepatocellular carcinoma (HCC) arise in patients with advanced liver disease, usually cirrhosis. Most patients with clinically evident HCC are not candidates for treatment with curative intent because of large tumor size, invasion of hepatic or portal veins, or metastatic disease. For this reason, screening for HCC at an asymptomatic and potentially curable stage in patients with advanced liver disease has been recommended by some authorities. Screening with various methods, of which ultrasound (US) and alpha-fetoprotein (AFP) have been the most extensively studied, has become accepted practice. Recently the technique of imaging the liver with or during both the hepatic arterial and portal venous phases of intravenous contrast ("liver-shuttle") has shown increased sensitivity in detecting HCCs compared to US.

The hypothesis of this study is that CT using a "liver-shuttle" protocol once a year is more sensitive and specific than US twice a year, both in combination with AFP for identification of potentially curable HCC in patients with cirrhosis. Patients will be randomized to "routine," accepted screening with hepatic US and AFP testing every 6 months or AFP testing every 6 months wtih triphasic CT every 12 months.

ELIGIBILITY:
Inclusion Criteria:

* liver biopsy or clinical diagnosis compatible with advanced liver fibrosis or cirrhosis
* potential candidate for treatment of HCC
* imaging study involving the liver in the last 12 months without evidence for HCC
* must be a veteran in VISN 23

Exclusion Criteria:

* active or untreated malignancy other than non-melanoma skin cancer
* patients with advanced medical conditions such as severe cardiovascular disease, COPD, or severe end-stage liver disease
* patients unable to receive intravenous contrast due to advanced kidney disease or severe allergy
* history of liver mass identified on imaging study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2001-11; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of screening measure to detect very early/early stage HCC (Barcelona Clinic Liver Cancer Staging System) | 6-12 months
  Confirmed diagnosis of hepatocellular carcinoma by biopsy or imaging according according to BCLC recommendations

SECONDARY OUTCOMES:
Cost - Effectiveness of screening measure | 1 year
  Cost of each screening protocol to identify one very early/early stage HCC

CONTACTS AND LOCATIONS:
Overall Officials: Christine Pocha, MD, PhD, Principal Investigator — Minneapolis Veterans Affairs Medical Center
Locations (1):
- Minneapolis Veterans Affairs Medical Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Pocha C, Dieperink E, McMaken KA, Knott A, Thuras P, Ho SB. Surveillance for hepatocellular cancer with ultrasonography vs. computed tomography -- a randomised study. Aliment Pharmacol Ther. 2013 Aug;38(3):303-12. doi: 10.1111/apt.12370. Epub 2013 Jun 10. PMID 23750991